CLINICAL TRIAL: NCT01002690
Title: Effect of COX-2 Inhibition on Allergen-induced Airway Obstruction in Subjects With Asthma
Brief Title: COX-2 Inhibition in Allergic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbro Dahlen (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Barbro Dahlen, MD PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: COX2EAR090531
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: Asthma; Allergen challenge; Airway responsiveness; Prostaglandins; Eicosanoids
MeSH Terms: conditions — Asthma | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etoricoxib (Experimental): 10-13 days treatment with etoricoxib
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Etoricoxib — 90 mg/day orally for 10-13 days
  Other Names: Arcoxia

SUMMARY:
The study is part of a research programme into mechanisms of asthmatic airway obstruction, focusing on the role of lipid mediators such as the prostaglandins.

To this end the effect of a non-steroidal anti-inflammatory drug, the selective COX-2 inhibitor etoricoxib, will be evaluated in the allergen challenge setting in twelve subjects with intermittent allergic asthma. Active treatment for 10 to 13 days will be compared with an identical study period with no treatment in a cross-over, randomised design. Rising dose allergen challenges will be performed on three occasions to assess possible changes in airways responsiveness. Sampling of blood, urine, saliva and sputum will be done to allow for analyses of the production of prostaglandins and other lipid mediators, of the efficacy of COX-2 inhibition as well as of regulation of immune cells.

It is hypothesized that inhibition of COX-2 by virtue of inhibition of bronchoprotective prostaglandin E2 leads to a slightly exaggerated airway response to allergen exposure.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 18 to 55 years inclusive
* A history of asthma for at least 6 months with at least one of the following:

  * response to standard asthma treatment
  * episodic wheezing
  * change in lung function over short periods of time
* A positive methacholine challenge test as evidenced by a PD20 ≤7256 µg cumulated dose within 8 weeks prior to screening or at the screening visit.
* Stable intermittent asthma, only using bronchodilator therapy as needed for the last 4 weeks.
* FEV1 ≥ 75% of predicted.
* A positive skin prick test to pollen (grass, birch, mugwort) or animal dander (dog, cat)

Exclusion Criteria:

* Known or suspected hypersensitivity to coxibs
* Any significant respiratory disease other than asthma
* Respiratory tract infection within 4 weeks before inclusion.
* Any significant disease or disorder which, in the opinion of the investigator, may put the patient at risk because of participation in the study. In particular previous or present history of cardiovascular disease, ie myocardial infarction, stroke, severe hypertension, left ventricular heart failure and/or pulmonary hypertension are strict exclusion criteria.
* Current or former smoker within the last year and a smoking history of >4 packyears
* Pregnancy/breastfeeding
* Use of:

  * inhaled glucocorticosteroid treatment or use of oral corticosteroids for the last 8 weeks prior to inclusion or during the study.
  * inhaled long-acting or oral beta2-agonists, anticholinergic bronchodilators, cromones, antihistamines, theophyllines and antileukotrienes within 2 weeks of screening or during the study.
  * paracetamol, NSAIDs or any other antiinflammatory drugs the last 2 weeks prior to inclusion or during the study.
  * need of any other regular drug treatment that may interfere with the study outcomes.
* BMI >30 kg/m2.
* Use of any beta-blocking agent
* Any non-asthma-related, clinically significant abnormal finding in physical and/or vital signs, and/or in hematology or blood chemistry tests at visit 1, which in the opinion of the investigator, may put the patient at risk because of participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Allergen PD20 FEV1 | 10 to 13 days

SECONDARY OUTCOMES:
Urinary prostaglandin E2 and D2 concentrations | 10-13 days

CONTACTS AND LOCATIONS:
Overall Officials: Barbro Dahlén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden